CLINICAL TRIAL: NCT06772948
Title: Effects of Telerehabilitation Based Clinical Pilates Exercises Applied to Health Care Workers With Problems of the Musculoskeletal System
Brief Title: Effects of Telerehabilitation-Based Clinical Pilates Exercises on Health Care Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUniver.
Record Dates: First submitted 2024-12-12; First posted 2025-01-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Healthcare Workers; Musculoskeletal Pain
Keywords: telerehabilitation; pilates; healthcare professionals; musculoskeletal system
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronised Group (Experimental): A six-week clinical Pilates exercise program will be applied to healthcare professionals via video conferencing (Zoom application) synchronized with a physiotherapist, for 40 minutes, two days a week.
  Interventions: Other: Synchronized group
- Asynchronised Group (Active Comparator): A six-week clinical Pilates exercise program will be applied asynchronously to healthcare professionals by watching videos on YouTube for 40 minutes, two days a week.
  Interventions: Other: Asynchronised group

INTERVENTIONS:
Other: Asynchronised group — Health workers with musculoskeletal system disorders will be given pilates exercises asynchronously using the YouTube application.
  Arms: Asynchronised Group
Other: Synchronized group — Using the Zoom application, healthcare workers with musculoskeletal disorders will perform pilates exercises synchronously.
  Arms: Synchronised Group

SUMMARY:
Musculoskeletal disorders can cause a decrease in employees' work continuity and job performance. During their working hours, healthcare workers stand for long periods of time, sit in wrong positions, actively use their upper extremities and work in incorrect postures. For this reason, they experience musculoskeletal system problems. This study was designed to determine the effectiveness of pilates exercises to be applied via tele-rehabilitation method for musculoskeletal system problems that may be seen in healthcare workers.

DETAILED DESCRIPTION:
Work-related disorders that can cause pain, limitation of movement and disability in working people and affect muscles, tendons and ligaments are called work-related musculoskeletal disorders (WMD). Work-related musculoskeletal disorders (WMSD) may occur acutely or chronically depending on age, occupation, activity level and lifestyle.

Health workers are people whose primary purpose is to take actions to improve health. They examine physical and mental problems, diagnose, treat and prevent problems based on the needs of the people they serve. It also conducts research and develops methods to improve evidence-based health services. Healthcare professionals include doctors, nurses, assistants, technicians, and assistants and provide care services to patients.

According to the European Union report, the number of work accidents in healthcare workers is 34% higher than in other professions.. In the 2012-2017 data of the Social Security Institution (SGK), 154 of 3040 occupational disease diagnoses (5.06%) consist of a musculoskeletal system disease. In a study, it was stated that the secondary diagnosis in healthcare workers was musculoskeletal system diseases, accounting for 15.2% (n = 17).In another systematic review examining the prevalence of musculoskeletal diseases in healthcare workers, the 1-year prevalence was found to be 28-96%. A study conducted by the American Nurses Association in 2011 showed that 56% of nurses experienced work-related musculoskeletal disorders.In a cross-sectional study conducted in Turkey in 2010, the 12-month prevalence was found to be 79.5%, and the highest prevalence was waist disorder (49.7%), followed by shoulder (38%) and neck (35%) disorders. A study investigating work-related BDSD in hospital employees found upper extremity pain during work in 58.1% of the employees. Other findings included stiffness, numbness, and swelling in the upper extremity. In another study, it was observed that IBD caused limitations in home and work activities, and an increase in the use of painkillers and the use of rest days in intensive care and operating room workers. In a study involving 78 midwives, at least one musculoskeletal system disorder was found in 67.6% of the participants. The highest prevalence was observed in the shoulder region with 44%, and the lowest prevalence was observed in the elbow (8%). A study investigating the relationship between physiotherapists' quality of life and physical activity level found physiotherapists to be one of the professional groups most prone to musculoskeletal problems.. In a study evaluating injury rates among physiotherapists, it was shown that 74% of physiotherapists working in the general physiotherapy department, 71% of physiotherapists working in the field of neurology, and 48% of physiotherapists working in the field of orthopedics had occupation-related musculoskeletal system problems. BDSRs in medical personnel and healthcare workers can cause difficulty in daily activities and leave work for nurses, nurse assistants, and hospital employees.Neck pain is the most common condition among nurses, and its 12-month prevalence was found to be 61.1%. Other risk areas for nurses were the lower back (47.2%), shoulders (46.7%), wrists and hands (27.3%) and elbow (13.9%). The most important reasons for the increase in upper extremity BDSR include being a woman, poor sleep quality, high physical activity level, poor ergonomics, increased workload and mental stress. In a study, the main reason for receiving a medical report among female hospital employees was found to be musculoskeletal disorders, and they determined that 28% of them required medical treatment.It is stated that low back pain is more common in women than men . They determined that the risk of pain is higher in women than in men and that body mass index is a risk factor that increases pain. Pain complaints increase in women with high body mass index. The risk of increased lower extremity pain is increased in obesity. According to World Health Organization estimates, 70-80% of deaths in developed countries and 40-50% of deaths in underdeveloped countries are caused by lifestyle-related diseases. Therefore, the health services to be provided should be aimed at protecting, maintaining and improving health. Healthcare professionals have important responsibilities in developing and maintaining these behaviors. That's why healthcare professionals must first correct their own lifestyle. When looking at the literature; In a study conducted to determine the healthy lifestyle behaviors of healthcare professionals, the lowest score was obtained from the exercise sub-dimension. In the study conducted to measure the health behaviors of healthcare personnel working in primary healthcare services, the lowest average score belongs to the exercise subfield (26). In a study conducted with nurses, it was stated that the rate of those who did not do physical activity was higher. In the study on health promotion behaviors of nursing school students, the lowest score was in the exercise sub-dimension. When the healthy lifestyle behaviors of healthcare professionals are examined according to their involvement in sports, the difference is significant and people interested in sports form healthy lifestyle behaviors better. Regular exercise has positive effects on health, such as weight control and cancer prevention. A suitable environment and time must be created for people to exercise regularly. It has been observed that healthcare workers who exercise 3-4 days a week or more get high scores on the Healthy Lifestyle Behaviors Scale (HLBD). However, since healthcare workers work on a shift system, they have difficulty in creating a suitable time and environment for exercise. Exercising via telerehabilitation may be an option that comes to mind in order to help healthcare professionals gain regular exercise habits and protect their health.

Telerehabilitation; It is a method that reduces service barriers such as time, cost and distance, and brings healthcare professionals and patients together in a virtual environment. Telerehabilitation enables the implementation of remote rehabilitation using technologies. Physiotherapists use telerehabilitation for evaluation, diagnosis, prognosis and treatment.

Pilates exercises were transferred to the clinic by Australian physiotherapists in the early 2000s and were called "clinical Pilates". The Clinical Pilates method is a mind-body exercise based on 6 principles: centering, concentration, control, precision, breathing and flow. Pilates exercises focus on spinal stabilization and are designed to build muscle strength, flexibility, balance, proprioception and body awareness. Breathing and muscle control during these exercises reduce pain and improve posture. The Clinical Pilates method can be applied as an exercise method for healthy people and sick people (10).Online Pilates exercises are an exercise that increases physical activity and provides positive effects in risky situations such as pandemics or when exercise centers cannot be reached.

When applying clinical pilates exercises, there are 5 elements that should be applied during the exercise. These; Breathing: Lateral breathing is used to maintain stabilization of the core muscles.

Centering: Central stabilization is achieved in the neutral spine position by activation of the Transversus abdominus, Pelvic floor muscles, and Multifidius.

Rib cage placement: The rib cage should be in a neutral position for correct muscle synergy and the neutral position should be maintained during extremity movements.

Shoulder Girdle Placement: Scapula-thoracic stabilization is achieved by activation of the rhomboid muscles, Serratus Anterior, and lower trapezius and is maintained throughout extremity movements.

Head-Neck Positioning: Without allowing the activation of the superficial neck flexors, the head-neck is placed in a neutral position and neck stabilization is achieved by activating the deep neck flexors.

A study has shown that online pilates exercises are almost as practical and easy to implement as face-to-face pilates exercises.

Healthcare workers may encounter risks and dangers due to their work areas and the normal order of work. In order to serve patients, they must first protect their own health.The aim of this study is to investigate the effectiveness of pilates exercises applied with two different tele-rehabilitation methods for the musculoskeletal system problems of healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* No health problems that prevent him from exercising
* Being between the ages of 25-50
* Lack of regular exercise habits
* Being a healthcare worker
* female gender
* Individuals with technological opportunities

Exclusion Criteria:

* Individuals who cannot participate in the exercise program regularly Individuals diagnosed with any orthopedic, neurological, rheumatological disease
* Individuals with pregnancy
* Individuals who follow a different exercise program

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 34 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Extended Nordic Musculoskeletal Questionnaire | through study completion, an average of 8 month
  The GNKİSA provides information on musculoskeletal pain in nine body regions (neck, shoulders, back, elbows, wrists/hands, waist, hips/thighs, knees, ankles/feet). . GNKISA asks about soreness, pain or discomfort in nine body regions so far, in the last 12 months, in the last four weeks and on the day of the assessment. The answer is yes/no and is filled in by the person or by interview technique.Turkish Validity and Reliability of the Questionnaire was made by in Kahraman et al.
Visual Analog Scale | through study completion, an average of 8 month
  The pain in the body part where the most pain is felt will be asked to be scored according to the Visual Analog Scale (VAS). VAS is used to evaluate pain and its severity on a scale of 0 - 10. The person being tested indicates the level of pain he/she feels using a straight horizontal line 10 cm long. The researcher then marks the indicated point. The range 0-3 indicates no or mild pain, the range 4-6 indicates severe pain, and the range 7-10 indicates very strong to the most severe pain
6 Minute Walk Test | through study completion, an average of 8 month
  6MWT involves walking back and forth as fast as possible along a 30 m straight path on a flat, hard surface for 6 minutes. The 6MWT duration is short, it is easy to perform, and the space required to perform the test.
Trunk Flexion Endurance Test | through study completion, an average of 8 month
  Participants will be placed in a sitting position with their hips and knees flexed at 90 degrees and their trunks at a 60-degree angle to the table, their backs are straight, their hands are crossed on opposite shoulders. The time the person maintains this position will be recorded.
Trunk Extension Endurance Test: | through study completion, an average of 8 month
  The participant's pelvis, knee and ankle will be fixed to the examination table and the participant will be positioned face down with the upper body extended over the edge of the table. The participant will be asked to remain in a horizontal position with arms crossed over the chest and the time spent in this position will be recorded.
Trunk Lateral Endurance Test | through study completion, an average of 8 month
  The participant will be asked to lift the hips by supporting the body with the feet while the elbow is in contact with the ground in a side-lying position.

SECONDARY OUTCOMES:
Flamingo Balance Test | through study completion, an average of 8 month
  People will be asked to balance by standing on their dominant foot on a wooden beam that is 50 cm long, 4 cm high and 3 cm wide, bending the other side's legs at the knee and holding the foot of this leg. People will be asked to try to stay in this position for 1 minute. When the balance is disturbed, the time will be stopped and when the balance is restored, the time will start. Each disturbance of balance will be recorded (34).
Sit-and-reach test | through study completion, an average of 8 month
  The person will be in a long sitting position on the floor with knees stretched and feet shoulder-width apart, and the soles of the feet will be in contact with the sit-and-reach table. The person will be asked to lean forward and forward. The difference between the first point and the last point will be measured with the ruler and recorded in cm.
Posture Analysis | through study completion, an average of 8 month
  A mobile application called "Posture:Al Medical Assistant" will be used to analyze the participants' posture. Photos of the participants will be taken from the front, back, right and left sides. Photos will be taken aligned according to the application's instructions. After taking the photo, body tilt, head, shoulders and hip tilt values will be reported in degrees by the application.
Waist-hip ratio | through study completion, an average of 8 month
  Waist-hip ratio will be checked to determine body composition. Waist circumference will be measured over the umbilicus and at the lowest rib level. Hip circumference will be measured with a tape measure from the widest area of the posterior hip. The ratio will be calculated with waist circumference is divided by hip circumference
Body mass index (BMI) | through study completion, an average of 8 month
  Weight will be calculated in kilograms, height will be measured in meters. BMI will be calculated by dividing the body weight in kilograms by the square of the height in meters.Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will share it to benefit future studies.
Supporting Information: Study Protocol, SAP
Time Frame: 10 November - 10 March

REFERENCES:
- [Background] Ou YK, Liu Y, Chang YP, Lee BO. Relationship between Musculoskeletal Disorders and Work Performance of Nursing Staff: A Comparison of Hospital Nursing Departments. Int J Environ Res Public Health. 2021 Jul 2;18(13):7085. doi: 10.3390/ijerph18137085. PMID 34281022
- [Background] Ross MH, Nelson M, Parravicini V, Weight M, Tyrrell R, Hartley N, Russell T. Staff perspectives on the key elements to successful rapid uptake of telerehabilitation in medium-sized public hospital physiotherapy departments. Physiother Res Int. 2023 Jul;28(3):e1991. doi: 10.1002/pri.1991. Epub 2022 Dec 20. PMID 36540908
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272
- [Background] Aloyuni S, Alharbi R, Kashoo F, Alqahtani M, Alanazi A, Alzhrani M, Ahmad M. Knowledge, Attitude, and Barriers to Telerehabilitation-Based Physical Therapy Practice in Saudi Arabia. Healthcare (Basel). 2020 Nov 4;8(4):460. doi: 10.3390/healthcare8040460. PMID 33158298
- [Background] Almhdawi KA, Alrabbaie H, Kanaan SF, Alahmar MR, Oteir AO, Mansour ZM, Obeidat DS. The prevalence of upper quadrants work-related musculoskeletal disorders and their predictors among registered nurses. Work. 2021;68(4):1035-1047. doi: 10.3233/WOR-213434. PMID 33867370